CLINICAL TRIAL: NCT05928910
Title: Decreasing Intraprocedural Peripheral Nerve Evaluation (PNE) Pain and Anxiety Using the SmileyScope Virtual Reality
Brief Title: Virtual Reality (VR) During Peripheral Nerve Evaluation (PNE) Procedure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decided to not proceed with study due to lack of personnel
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Raveen Syan, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230398
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SmileyScope VR Group (Experimental): Participants in this group will wear the SmileyScope VR set during the PNE procedure for approximately 40 minutes.
  Interventions: Device: SmileyScope VR
- No VR Group (Experimental): Participants in this group will receive standard of care treatment.
  Interventions: Other: Standard of Care Treatment

INTERVENTIONS:
Device: SmileyScope VR — The SmileyScope Virtual Reality Headset is a VR headset to reduce pain and anxiety undergoing medical procedures. The device comes pre-loaded with a static virtual reality scenario. Participants will use the device in person when coming to clinic during an in-person, one time PNE procedure.
  Arms: SmileyScope VR Group
Other: Standard of Care Treatment — Participants in this group will receive standard of care treatment during an in-person, one time PNE procedure.
  Arms: No VR Group

SUMMARY:
The purpose of this research is to evaluate whether or not wearing a virtual reality headset affects pain and anxiety in patients undergoing percutaneous nerve evaluation (PNE).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective peripheral nerve evaluation studies for pelvic floor dysfunction

Exclusion Criteria:

* Have a serious comorbid illness or condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study
* Significant refractive error, unilateral blindness, epilepsy, or other conditions such as skin infections, cancers, etc., which could compromise the physical function of the headset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change In Pain as Measured by Numeric Pain Scale | Baseline (pre-PNE procedure), up to 1 hour (post-PNE procedure)
  Pain will be measured using the numeric pain scale. Scores range from 0-10. Higher scores indicate worse pain.
Change in Anxiety as Measured by State Trait Anxiety Inventory | Baseline (pre-PNE procedure), up to 1 hour (post-PNE procedure)
  Anxiety will be measured using the State Trait Anxiety Inventory. Scores range from 0-24. Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
Satisfaction with Procedure as measured by Likert Scale | up to one hour post-procedure
  Satisfaction with be measured by likert scale. Scores range from (1) very unsatisfied with today's procedure to (5) very satisfied with today's procedure.
Feasibility for the Utilization of the Smiley Scope VR Headset by Likert Scale | up to one hour post-procedure
  Feasibility will be measured by a 5-point Likert scale for the utilization of the Smiley Scope VR Headset. Scores range from (1) very unhelpful in managing your pain and anxiety associated with the PNE procedure to (5) very helpful in managing your pain and anxiety associated with the PNE procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Raveen Syan, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No